CLINICAL TRIAL: NCT01362218
Title: Cardiovascular Fixed Combination Pill ASR: Pharmacodynamic Clinical Trial of a Fixed Dose Combination of Acetylsalicylic Acid, Simvastatin, and Ramipril (Cardiovascular Polypill); LDL Cholesterol
Brief Title: Pharmacodynamic Clinical Trial of Cardiovascular Polypill on LDL Cholesterol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per sponsor's decision
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P-100820-01
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Elevated LDL Cholesterol
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Blood Circulation; Aspirin; Simvastatin; Ramipril

ARMS (2):
- Fixed Dose Combination Pill (Experimental): A fixed dose combination of acetylsalicylic acid, simvastatin, and ramipril Intervention: Drug: Cardiovascular fixed dose combination pill (acetylsalicylic acid, simvastatin and ramipril)
  Interventions: Drug: Cardiovascular fixed dose combination pill (acetylsalicylic acid, simvastatin and ramipril)
- Simvastatin (Active Comparator): Simvastatin given together with the reference drugs ramipril and acetylsalicylic acid
  Interventions: Drug: Simvastatin, ramipril, acetylsalicylic acid

INTERVENTIONS:
Drug: Cardiovascular fixed dose combination pill (acetylsalicylic acid, simvastatin and ramipril) — A once daily oral dose of the cardiovascular fixed dose combination pill ( acetylsalicylic acid, simvastatin, ramipril) for 8 weeks.
  Arms: Fixed Dose Combination Pill
Drug: Simvastatin, ramipril, acetylsalicylic acid — A once daily oral dose of simvastatin, ramipril, acetylsalicylic acid for 8 weeks
  Arms: Simvastatin

SUMMARY:
This study evaluates the effect on LDL cholesterol of the 3 drugs given together in the cardiovascular fixed dose combination pill (acetylsalicylic acid, simvastatin, and ramipril) as compared to the effect on LDL cholesterol of the reference products (simvastatin, ramipril, acetylsalicylic acid) Approximately 350 subjects will be screened, 266 randomized in order about 238 subjects to finish the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 and <75 years.
* Previously untreated or not treated with fibrates during the last 6 weeks or with any other lipid lowering drug for the last 4 weeks.
* LDL-cholesterol ≥130 and ≤220 mg/dL.
* Systolic blood pressure ≥120 and <160 mmHg and diastolic blood pressure ≥70 and <100 mmHg.
* Provide written informed consent.

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difference in LDL-cholesterol levels between the basal and the final visit of treatment period. | Day 56

SECONDARY OUTCOMES:
• Difference in VLDL-cholesterol levels between the basal and the final visit of treatment period. | Day 56
• Difference in HDL-cholesterol levels between the basal and the final visit of treatment period. | Day 56
• Difference in total cholesterol levels between the basal and the final visit of treatment period. | Day 56
• Difference in triglyceride levels between the basal and the final visit of treatment period | Day 56

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain